# The Feasibility of the VOICES Digital Health Tool for Elder Mistreatment Screening in the Primary Care Setting

(VOICES-PC Feasibility)

Protocol Number 2000031059 Protocol Version 01/20/2022 Version #1.01

#### PRINCIPAL INVESTIGATOR:

Fuad Abujarad
Yale School of Medicine
Department of Emergency Medicine
(203)928-9259
Fuad.abujarad@yale.edu

**Confidentiality Statement:** 

## **REVISION HISTORY:**

| Revision # | Version Date |
|------------|--------------|

# **Synopsis**

## **Primary Objective**

The primary objective of this study is to perform a feasibility evaluation of the VOICES screening tool (HIC#: 2000023799) among 80 older adults in primary care settings.

#### Secondary Objective (if applicable)

#### **Study Duration**

Approximately 10 months.

#### Study Design

This is a feasibility study of a tablet-based screening tool to identify suspicion of elder mistreatment.

#### **Number of Study Sites**

1: Yale Internal Medicine Associates (YIMA).

#### **Study Population**

Older adults (age 60+) seen at YIMA.

#### **Number of Participants**

80

#### **Primary Outcome Variables**

Feasibility and Acceptability

#### **Secondary and Exploratory Outcome Variables (if applicable)**

N/A

# **Abbreviations**

| Abbreviation | Explanation |
|--------------|-------------------------------------------------|
| ЕМ | Elder Mistreatment |
| YIMA | Yale Internal Medicine Associates |
| PSE | Connecticut Protective Services for the Elderly |
| RA | Research assistant |
| PC | Primary Care |

#2000031059

# **Glossary of Terms**

| Glossary | Explanation |
|----------|-------------|
|----------|-------------|

# **Table of Contents**

| Pr | reface | | 2 |
|----|--------|---------------------------------------------------------|----|
| Sy | ynopsi | S | 4 |
| | Prima | ry Objective | 4 |
| | Secor | ndary Objective (if applicable) | 4 |
| | Study | Duration | 4 |
| | Study | Design | 4 |
| | Numb | per of Study Sites | 4 |
| | Study | Population | 5 |
| | Numb | per of Participants | 5 |
| | Prima | ry Outcome Variables | 5 |
| | Secor | ndary and Exploratory Outcome Variables (if applicable) | 5 |
| Αŀ | bbrevi | ations | 6 |
| G | lossar | y of Terms | 7 |
| 1 | Intr | oduction | 11 |
| | 1.1 | Introductory Statement | 11 |
| 2 | Bac | ckground | 12 |
| | 2.1. | .1 Device Preclinical Experience | 12 |
| | 2.1. | .2 Device Clinical Experience | 12 |
| | 2.2 | Background/prevalence of research topic | 12 |
| 3 | Rat | ionale/Significance | 13 |
| | 3.1 | Problem Statement | 13 |
| | 3.2 | Purpose of Study/Potential Impact | 13 |
| | 3.2 | .1 Potential Risks | 13 |
| | 3.2 | .2 Potential Benefits | 13 |
| 4 | Stu | dy Objectives | 14 |
| | 4.1 | Hypothesis | 14 |
| | 4.2 | Primary Objective | 14 |
| | 4.3 | Secondary Objectives (if applicable) | 14 |
| 5 | Stu | dy Design | 15 |
| | 5.1 | General Design Description | 15 |

| | 5.1.1 | Study Date Range and Duration | 15 |
|---|---|---|---|
| | 5.1.2 | Number of Study Sites | 15 |
| | 5.2 | Outcome Variables | 15 |
| | 5.2.1 | Primary Outcome Variables | 15 |
| | 5.2.2 | Secondary and Exploratory Outcome Variables (if applicable) | 15 |
| | 5.3 S | tudy Population | 15 |
| | 5.3.1 | Number of Participants | 16 |
| | 5.3.2 | Eligibility Criteria/Vulnerable Populations | 16 |
| 6 | Metho | ods | 19 |
| | 6.1 T | reatment – Device | 19 |
| | 6.1.1<br>being | Intended Use for Device (provide the following information for each device investigated in the study) | |
| | 6.1.2 | Device Administration and Schedule | 19 |
| | 6.1.3 | Method of Assignment/Randomization (if applicable) | 19 |
| | 6.1.4 | Device Calibration | 19 |
| | 6.1.5 | Storage Conditions | 19 |
| | 6.1.6 | Concomitant therapy | 19 |
| | 6.1.7 | Restrictions | 19 |
| | 6.2 A | ssessments | 20 |
| | 6.2.1 | Efficacy | 20 |
| | 6.2.2 | Safety | 20 |
| | 6.2.3 | Adverse Events Definition and Reporting | 21 |
| | 6.2.4 | Pharmacokinetics (if applicable) | 21 |
| | 6.2.5 | Biomarkers (if applicable) | 21 |
| | 6.3 S | tudy Procedures | 21 |
| | 6.3.1 | Study Schedule | 22 |
| | 6.3.2 | Informed Consent | 22 |
| | 6.3.3 | Screening | 22 |
| | 6.3.4 | Enrollment | 22 |
| | 6.3.5 | On Study Visits | 22 |
| | 6.3.6 | End of Study and Follow-up | 23 |
| | 6.3.7 | Removal of subjects | 23 |

| | 6.4 | Statistical Method | 23 |
|---|---|---|---|
| | 6.4. | 1 Statistical Design | 23 |
| | 6.4. | 2 Sample Size Considerations | 23 |
| | 6.4. | 3 Planned Analysis | 23 |
| | 6.4. | 4 Subsets and Covariates | 24 |
| | 6.4. | 5 Handling of Missing Data | 24 |
| 7 | Tria | I Administration | 25 |
| | 7.1 | Ethical Considerations: Informed Consent/Assent and HIPAA Authorization | 25 |
| | 7.2 | Institutional Review Board (IRB) Review | 25 |
| | 7.3 | Subject Confidentiality | 25 |
| | 7.4 | Deviations/Unanticipated Problems | 26 |
| | 7.5 | Data Collection | 26 |
| | 7.6 | Data Quality Assurance | 26 |
| | 7.7 | Study Records | 26 |
| | 7.8 | Access to Source | 26 |
| | 7.9 | Data or Specimen Storage/Security | 27 |
| | 7.10 | Retention of Records | 27 |
| | 7.11 | Study Monitoring | 27 |
| | 7.12 | Data Safety Monitoring Plan | 27 |
| | 7.13 | Study Modification | 27 |
| | 7.14 | Study Discontinuation | 27 |
| | 7.15 | Study Completion | 28 |
| | 7.16 | Conflict of Interest Policy | 28 |
| | 7.17 | Funding Source | 28 |
| | 7.18 | Publication Plan | 28 |
| 8 | App | endices | 29 |
| a | l iet | of Tables | 30 |

# 1 Introduction

## 1.1 Introductory Statement

This document is a protocol for a human research study. The purpose of this protocol is to ensure that this study is to be conducted according to ICH GCP guidelines, and according to CFR 21 Part 812, other applicable government regulations, and Institutional research policies and procedures.

# 2 Background

#### 2.1.1 Device Preclinical Experience

The VOICES tool has been developed and tested with more than 800 patients at Yale Emergency Department (IRB Protocol ID:2000023799 and Submission ID:CR00008317).

#### 2.1.2 Device Clinical Experience

In a prior clinical study at Yale Emergency Department (IRB Protocol ID:2000023799 and Submission ID:CR00008317), we developed an innovative digital health tool that runs on tablets called **VOICES** that screens, educates, and motivates older adults to make an informed decision about self-reporting of elder mistreatment. The **VOICES** tool is currently being evaluated with older adults *in emergency department settings*. *More than* 800 older adults have used the VOICES tool so far without any issues. Study participants have demonstrated signs of feasibility, acceptance, demand, and full completion of the tool for those who consented to participate. There is an opportunity to expand the use of the **VOICES** tool to a more vulnerable older adult populations, such as older adults in primary care settings.

#### 2.2 Background/Prevalence of Research Topic

Elder mistreatment (EM) is a major public health problem with estimated prevalence in the United State ranges from 27.9% to 62.3% for emotional abuse and 3.5%–23.1% for physical abuse among older adults with cognitive impairment (CI). EM consists of physical, emotional, sexual and financial abuse as well as neglect committed by a person in a position of trust to the older adult. It causes serious adverse outcomes for its victims including injury, increased service utilization, mental distress and the risk of mortality. A major barrier in overcoming EM is the inability to accurately identify EM victims. It is estimated that only 1 in 24 cases become known to authorities.

There are several perceived barriers to self-disclosure (informing others about the EM experiences) that limit help-seeking behaviors, including fear of nursing home placement, of losing autonomy or a caregiver, and of getting an abusive family member in legal trouble. As a result, reporting of EM remains low and providers often miss the opportunity to identify EM at point-of-care.

In our parent project, we used Digital Health frameworks to develop the Virtual cOaching in making Informed Choices on Elder Mistreatment Self-Disclosure (VOICES) tool. This is a new and innovative digital health tool that screens, educates, and motivates older adults to make an informed decision about self-identification (recognizing that they themselves are victims) and self-disclosure of elder mistreatment.

# 3 Rationale/Significance

#### 3.1 Problem Statement

Is the VOICES tool (IRB Protocol ID:2000023799 and Submission ID:CR00008317), currently developed for older adults and evaluated in emergency department settings, feasible for use for older adults in primary care settings?

#### 3.2 Purpose of Study/Potential Impact

Our aim is to perform a feasibility evaluation (N=80) of the VOICES screening tool among older adults in the primary care setting. If VOICES is feasible for identifying suspicion of EM in primary care setting, then we will be able to connect more victims of EM to necessary services and potentially prevent a multitude of poor EM outcomes.

#### 3.2.1 Potential Risks

There are no medical interventions in this study, and direct medical risks are minimal. However, identification of potential EM without adequate safeguards could increase the risk of physical harm, emotional harm, risk of neglect, and financial loss to the victim. In addition, EM identification can potentially lead to adverse events including:

- retaliation of a family member or caregiver,
- an older adult may lose the caregiver or be abandoned by a caregiver, and a family member or paid caregiver may be arrested / incarcerated,
- discharge of a patient to a long-term care or skilled nursing facility, which they
  may not be able to afford,
- distress/anxiety during and/or after using the VOICES tool is a potential risk given the complex emotions typically associated with this phenomenon.
- there is a risk of compromised security of personal information.

Many of these adverse events would likely occur as a result of the mandatory report to Connecticut Protective Services for the Elderly (PSE) that the care team (case manager, clinician, nurses, and attendings) would make. However, during this study the care team is NOT expected to discover information that will require them to make a report to PSE.

#### **Minimizing Risks:**

Risks will be minimized through appropriate participant exclusions and close medical supervision throughout the protocol. We will inform all participants that there is a chance that they may experience adverse events due to the identification of EM by participating in the study and that their participation is voluntary. We will also remind participants that they can discontinue participation at any time.

In Summary: VOICES' goal is to help identify cases of EM. The subsequent procedures for the EM identification are important but are similar to the case when a provider identify suspicion of EM during normal clinical care:

- all patients who screen positive with the VOICES tool will be reviewed and assessed by YIMA care team.
- while the research team recognizes that the EM identified through the VOICES tool may lead to risks for patients that are usually associated with EM identification, we anticipate that the care team response will minimize the possible adverse events due to the EM identification.
- We will train all RAs to detect common signs of distress and anxiety. If any are even suspected of being observed, the care team at YIMA, will be contacted immediately for consultation and next steps, which could include counseling, referrals, or a psychiatric evaluation.
- If the older adult screens positive on the VOICES for EM or the older adult
  wants to self-disclose EM, the RA will notify the care team in the YIMA that
  there is suspicion of EM. Also, if the tool fails to identify EM but the patient
  would like to disclose EM, the RA will notify the care team. The RA will stay
  with the participant until a member of the care team arrives and implements
  existing protocols for handling EM identification.

- The care team can address each patient's concerns around reporting, immediate safety concerns, and any concerns for retaliation or abandonment. If the assessment indicates suspicion of abuse, and the case gets reported to PSE, usually PSE will arrive within 12 hours to take care of the case. While waiting for PSE, the health care team members will discuss safety issues with the patient.
- We will protect against psychological distress by informing all participants that there is a chance that they may experience some negative emotions while completing the surveys, after completing survey, or when they leave the hospital, but that they do not have to answer questions that they find distressing. We will also remind participants that they can discontinue participation at any time. We will also provide all older adults that we approach with the brochure on resources for aging well that also include free referral line. These options will be discussed with participants during initial recruitment.
- Although privacy and confidentiality will be preserved to the utmost extent possible, participants will be informed that, should EM be identified, the RA will report this to the care team in the YIMA. For example, if in the course of research procedures, a participant reveals elder abuse to the RA, the RA will discuss with the participant his/her responsibility to report the abuse to the care team. The physician will be notified of any suspicion of abuse and will determine through an evaluation whether the patient is in immediate danger or requires a report to PSE. If the care team performs the EM assessment and finds a suspicion of abuse, they will intervene to ensure patient safety. Also, if the participant divulges suicidality, the RA must report this to the care team and notify the PI.
- We will follow standard hospital operating procedures to guard against the
  possibility of study coercion, loss of confidentiality, psychological distress, and
  escalation of abuse, acknowledging that awareness or suspicion of reporting
  may anger the abuser but can also empower the patients and ultimately, make
  them safer.
- Our intent is to conduct a VOICES study session without the presence of the caregiver/LAR. From our experience, family members usually volunteer to leave the room.
- We will ask the caregivers to leave the room before engaging the older adults in using the VOICES tool and after the consent and assent. If the older adult wants the caregiver to remain, we will respect their wishes, but that patient will be excluded from the study and no study information will be presented.
- If a participant reveals depression, the research assistant will notify the care team. If a participant reveals severe depression or suicidality, or requests immediate psychiatric care for any reason, the RA will alert the patient's clinician to initiate an immediate psychiatric evaluation.
- Since the VOICES tool is a web-based application in nature, **no information** will be stored on the tablet. If the tablet gets lost or stolen, the patient's data

#2000031059

01/20/22 Version #1.01

will not be compromised. All iPads contain encryption software, per University Policy 5100.

#### 3.2.2 Potential Benefits

Although there are risks to the subjects, the benefits outweigh the risks. EM can have profound medical consequences for victims, significantly increasing their risk for mortality, exacerbations of chronic illnesses, and depression. EM is very seldom identified, and low rates of identification and reporting have likely led to much of the associated morbidity and mortality. Therefore, by increasing identification of this morbid and mortal phenomenon, the VOICES tool may offer significant benefits to patients. A potential benefit for the participants is that they will gain better self-awareness, enhance and support self-disclosure, and improve reporting of EM at the point-of-care setting, which may result in, better emotional and physical health, increased safety, and quality of care.

# 4 Study Objectives

## 4.1 Hypothesis

The hypothesis of this study is: the VOICES tool, developed for older adults in emergency department settings, will be applicable and feasible for older adults in primary care settings?

- To what extent is VOICES likely to be used?
- To what extent is VOICES usable for end-users?
- To what extent is VOICES acceptable to end-users?
- To what extent can VOICES be delivered to participants in the context of the YIMA?
- To what extent can VOICES be carried out with older adults without outside intervention?

#### 4.2 Primary Objective

The primary objective of this study is to determine whether VOICES tool is feasible for identifying suspicion of elder mistreatment among older adults in primary care settings.

#### 4.3 Secondary Objectives (if applicable)

N/A.

# 5 Study Design

## 5.1 General Design Description

**Overview and Rationale:** We will conduct a feasibility evaluation (N=80) of the VOICES screening tool among older adults. *The objective of this study is to evaluate* feasibility *of the tool to guide modification and enhancement of the VOICES tool for use in the future pilot study.* 

**Settings:** Participants for the feasibility evaluation will be recruited from the large and diverse patient population that visit the YIMA.

**Sample Size Justification:** We will recruit eighty participants (N=80) from YIMA, targeting older adults age 60+ from diverse racial and ethnic backgrounds.

Our goal is to enroll enough subjects to identify themes, issues, and patterns related to feasibility. We anticipate some participants may not be able to use VOICES to completion.

**Recruitment:** The one-on-one evaluation sessions will last 45-60 minutes, and the method of conducting a single study session is as follows:

#### 5.1.1 Study Date Range and Duration

The expected length of the study is 45-60 minutes, will be completed in one session following consent of the individual and there will be no follow-up.

## 5.1.2 Number of Study Sites

This study will be performed at one study site, the YIMA.

#### 5.2 Outcome Variables

#### 5.2.1 Primary Outcome Variables

The primary outcome variables include the areas of feasibility of the VOICES tool.

- Usability: To what extend is VOICES usable to end-users?
- Acceptability: To what extent is VOICES satisfying to end-users?
- Demand: To what extent is VOICES likely to be used?
- **Implementation:** To what extent can VOICES be delivered to participants in the defined, context of the YIMA?
- **Practicality:** To what extent can VOICES be carried out with intended participants without outside intervention?

#### 5.2.2 Secondary and Exploratory Outcome Variables (if applicable)

N/A

#### 5.3 Study Population

Participants without cognitive impairment aged 60 and older seen at YIMA.

#### 5.3.1 Number of Participants

The number participants to be recruited is 80 participants.

#### 5.3.2 Eligibility Criteria/Vulnerable Populations

#2000031059

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

- 1. Age 60 or above
- 2. Living in Community Dwelling
- 3. Able to consent and communicate in English
- 4. Has no risk of COVID-19
- 5. Agrees and able to use the iPad
- 6. Stated willingness to comply with all study procedures and availability for the duration of the study
- 7. Provision of signed informed consent, or assent if LAR provides consent

An individual who meets any of the following criteria will be excluded from participation in this study:

- 1. Subjects who live in nursing homes or other long-term care setting
- 2. At the discretion of the clinician, patient will be excluded if they cannot safely undergo the studies required for participation
- 3. Patient refusal to participate
- 4. Severe cognitive, hearing, or vision impairment

# 6 Methods

#### 6.1 Treatment - Device

# 6.1.1 Intended Use for Device (provide the following information for each device being investigated in the study)

The VOICES tool is intended to be used primarily to identify suspicion of elder mistreatment.

#### 6.1.2 Device Administration and Schedule

The VOICES tool will be provided on an iPad to the eligible participant and self-administrated by the participant. The research assistant will provide technical assistance if necessary, but otherwise the participant is expected to go through the tool independently, guided by the tool's virtual coach.

We will assess the patient ability to consent by checking if the patient can:

- articulate a choice regarding study participation
- understand its purpose
- comprehend that participation does not constitute medical treatment

If the patient has the capacity to consent, then he/she will complete the consent process on their own.

If patient does not have the capacity to consent, the LAR will need to consent.

If the LAR is not present at the clinic, we will seek to obtain the consent remotely.

After the patient completes the consent process and (if needed) the LAR completes the consent process, the LAR will be asked to wait in the waiting room and away from the room where study is being conducted. The patient will undergo the study procedures on their own without the presence of the LAR. If the LAR did not leave the room, or if the patient wanted them to be present then the patient will not be eligible for the study and cannot participate.

## 6.1.3 Method of Assignment/Randomization (if applicable)

N/A

#### 6.1.4 Device Calibration

N/A

#### 6.1.5 Storage Conditions

All tablets will be secured in a locked cabinet when not in use.

#### 6.1.6 Concomitant therapy

NA

#### 6.1.7 Restrictions

N/A

#### 6.2 Assessments

#### 6.2.1 Efficacy

Questionnaires/metrics to be administered:

- Demographics questionnaire
- Post-Use Exit Survey questionnaire
- Verbal feedback

Demographics will be used to confirm the recruitment of a diverse population, as well as identify any patterns in outcomes with certain populations. The post-use exit survey will be used to determine some measures in feasibility.

#### 6.2.2 Safety

All data will be entered into databases that are protected with appropriate passwords and routine backups of all data will be carried out. All data collected on the subjects will be coded with numbers to maintain confidentiality. Access to the files will be restricted to the investigators and study personnel on this protocol. Clinical data will be stored with specific patient identifiers, (de-identification of samples), and maintained in a locked file, separate from any other clinical records with limited access, to assure patient confidentiality. Results will be assembled with confidential clinical research records, but will be unidentifiable without these files, to assure confidentiality. The only data that will be used in this study is the information directly obtained from the subjects.

#### 6.2.3 Adverse Events Definition and Reporting

An adverse event that must be reported to the IRB because it is one of the following:

- 1. Serious or life-threatening; AND
- 2. Unanticipated (unexpected) OR anticipated but occurring with a greater frequency than expected; AND
- 3. Possibly, probably or definitely related to the intervention.

This section describes the procedures and timelines for adverse events (AE) and serious adverse events (SAE), collection and reporting.

- No SAEs are expected from the direct use of VOICES tool on the iPad, but when SAEs occur as result of EM identification and disclosure that are related to the VOICES tool, they will be reported to the Yale IRB, and to the research team within 48 hours of study's knowledge of the SAE.
- AEs will be reported per Yale IRB policies. They will also be reported to the study's team. At minimum, included in semi-annual reports.
- In the unlikely event that such events occur, Reportable Events (which are events
  that are serious or life-threatening and unanticipated and possibly related)or
  Unanticipated Problems Involving Risks to Subjects or Others (UPIRSOs) that may
  require a temporary or permanent interruption of study activities will be reported
  immediately to the Yale IRB, and to the research team, followed by a written report
  within 5 calendar days of the Principal Investigator becoming aware of the event to
  the IRB and any appropriate funding and regulatory agencies.
- The PI will apprise fellow investigators and study personnel of all UPIRSOs and adverse events that occur during the conduct of this research project through regular study meetings and via email as they are reviewed by the PI.
- All deaths will be reported within 24 hours of study's knowledge of death.
- The report of death will be submitted to Yale IRB, and to the research team.
- Since the VOICES tool is a web-based application in nature, no information will be stored on the tablet. Data will be stored on Yale's secure servers. If the tablet becomes lost or stolen, the patient's data will not be compromised. All iPads contain encryption software, per University Policy 5100.

#### 6.2.4 Pharmacokinetics (if applicable)

N/A

#### 6.2.5 Biomarkers (if applicable)

N/A

## 6.3 Study Procedures

#### 6.3.1 Study Schedule

Only one visit and no follow-up. The study will be carried out in one session, during the duration of the participant's visit in the YIMA setting. There will be no follow-up with the participant, and the expected time to perform the study is around 45-60 minutes, including consent and post-use survey.

#### 6.3.2 Informed Consent

We will pay special attention to the ethical issues and the unique challenges of EM research as well as to consenting and enrolling older persons in our study. The consent process informs a volunteer about the study and fully explains the purpose of the research, that this is a research study, that participation is voluntary, and that the participant has the right to stop at any time. Our consent includes all of the eight basic elements of informed consent as articulated by 45 CFR §46.116,21 CFR §50 and Yale IRB Policy 200 Informed Consent for Human Research) and the additional elements of informed consent. Before agreeing to participate in VOICES, potential subjects (and if needed their LAR) will be made aware of and understand the risks of participation. They are the following:

- A statement that the study involves research. This includes:
  - An explanation of the purposes of the research, stressing that this is not an intervention
  - The expected duration of the subject's participation
  - A description of the procedures to be followed
  - A description of any foreseeable risks or discomforts to the subject.
  - A description of any expected benefits to the subject or to others
  - o When applicable, a disclosure of appropriate alternative
  - o A statement explaining how confidentiality of data will be managed
  - An explanation of the risk of injury
  - List of whom to contact with questions about the research, research subjects' rights, or in the event of a research-related injury to the subject, that include: Principal Investigator's contact information and IRB Administrator's contact information
- A statement that:
  - Participation is voluntary
  - Refusal to participate will involve no penalty or loss of benefits to which the subject is otherwise entitled
  - The subject may discontinue participation at any time without penalty or loss of benefits to which the subject is otherwise entitled.
- In addition to the eight required elements of informed consent, additional elements are added to the consent. They include:
  - A statement that VOICES may involve risks to the subject which are currently unforeseeable:

- Anticipated circumstances in which the subject's participation may be terminated by the PI;
- Any additional costs to the subject that may result from participation in the research;
- The consequences of a subject's decision to withdraw from the research and procedures for orderly termination of participation by the subject;
- o The approximate number of subjects involved in the study;
- An explanation of what will be done with the participant information, in the presenting case as well as long-term.

At the end of the consent process, the RA will review the subject's understanding of the study by asking the following question:

- o What are you being asked to do?
- O What questions is this study trying to answer?
- What are the potential risks and benefits of participating in this study?
- Can you withdraw from the study, and what should you do if you decide to withdraw?
- Do you understand that participation in this study is voluntary and is not part of your medical treatment?

#### 6.3.3 Screening

The study RA will be stationed in the YIMA and will work with designated YIMA personnel to identify potential participants.

- The research assistant (RA) will work with the case managers at the YIMA to identify
  potential participants among the already scheduled visits to the YIMA for the
  upcoming few weeks. YIMA staff may call eligible patients ahead of their upcoming visit
  to briefly introduce the study and determine if the older adult would like to participate to
  provide advance notice of the study.
- When a potential participant is identified, the front disk, RA, or the care team will
  contact the older adult or the Legally Authorized Representative (LAR) and inform
  them that they might be eligible to participate in an ongoing study. If they are
  interested, then they will need to account for an extra 45-60 minutes during their visit
  to YIMA.
- The RA will be stationed in the YIMA and will work with designated case manager to identify potential participants during their regular visit to the YIMA.

We are requesting a HIPPA waiver for recruitment purposes only. The RA will work with case manager and will review the EPIC screen and will then check the demographic for patient 60 years or older. The case managers will help the RA approach the patients to ask additional screening questions. We don't have resources and staffing to approach every **YIMA** patient and ascertain eligibility. Using Epic is more efficient for the RAs. The RA will track and document each EHR that the RA accesses using the VOICES tool screening log.

#### 6.3.4 Enrollment

- The YIMA staff will approach the patients at the YIMA and introduce the study and the RA. If the older adult wants to participate, the RA will conduct eligibility screening.
- The RA will enroll subjects in the study, after they have consented and meet all eligibility criteria.

#### 6.3.5 On Study Visits

There will be only one study visit necessary, which will be approximately a 45–60-minute session including:

- Introduction of study by research assistant
- Consent/Assent
- VOICES Tool self-administered by the eligible subject
- Post-use survey
- Incentive and resources to be given at end of study
- If the patient is eligible and would like to participate in the study, the RA will conduct the consent process (and if needed a consent from the LAR and assent from the subject) in a private exam room dedicated for this study. Participants (and if needed their LAR) must be able to consent and communicate in English. For all patients participating in this study, the consent will be requested from the patient and if needed from the LAR. Participants must be able and agree to use a tablet computer.
- If the LAR is needed for consent, and present in the clinic, verbal consent will be obtained.
- If the LAR is needed for consent and is not present in the clinic, verbal consent will be obtained via telephone.
- Important considerations
  - At the end of the consent process, the RA will review the subject's understanding of the study by asking the following question:
    - O What are you being asked to do?
    - o What questions is this study trying to answer?
    - What are the potential risks and benefits of participating in this study?
    - Can you withdraw from the study, and what should you do if you decide to withdraw?
    - Do you understand that participation in this study is voluntary and is not part of your medical treatment?
  - The caregiver ( if any is present ) will be asked to step out of the room and go wait in the family room. The patient will undergo the study producers on their own without the presence of the caregiver. If the caregiver did not leave the room, or if the patient wanted them to be present then the patient will not be eligible for the study and cannot participate.
  - Participants will be given a description of the study and that they are testing the feasibility of VOICES and that the evaluation is not a measure of their individual performance but measure of the tool performance.
  - The RA will collect the participant demographics to gather background information on the participants.

- Participants will be asked to go through the VOICES tool to completion, when
  possible, and to think aloud, verbalizing any confusion while performing tasks, in
  order to identify areas of difficulty when performing the tasks. The RA will be
  monitoring the use of VOICES and documenting issues of interest that are observed.
- The RA will collect the post study survey from participants after using VOICES.
- Each participant will be given \$75 Bank of America gift card as compensation for their time and participation.
- If participant screen positive or want to self-report EM, the RA will notify the care team
- The RA will stay with the older adult until a member of the care team comes.

#### 6.3.6 End of Study and Follow-up

Participants will be given a \$75 incentive upon completion of the post-use survey, as well as a brochure on resources from the CT Protective Services for the Elderly. There will be no follow-up visits or contact required from the participant, and any data gathered from the participant up until their withdrawal will continue to be used for data analysis purposes.

#### 6.3.7 Removal of subjects

Since this study is a one-time study, if a participant decides to withdraw, the participant's withdrawal will be documented in the study record and the study will not continue from the point of their withdrawal. Also, the participant will be told that they can quit the study at any time.

#### 6.4 Statistical Method

#### 6.4.1 Statistical Design

The purpose of this objective is to understand important areas of feasibility. Data for the completion of this objective comes from the following sources: (1) Participant demographic data obtained on pre-survey, (2) participant verbal feedback given to RA (3) participant responses given to questions on post-survey, and (4) observations made by the RA on enrollment, VOICES administration, and data collection for each participant.

#### 6.4.2 Sample Size Considerations

**Sample Size Justification:** We will recruit twenty participants (N=80) from the YIMA over a 8-month period. We will target older adults age 60+ from diverse racial and ethnic backgrounds. Our goal is to identify themes, issues, and patterns related to feasibility. We anticipate some participants may not be able to use VOICES to completion.

#### 6.4.3 Planned Analysis

#### 6.4.3.1 Primary Analyses

Data analysis will be performed using SAS v9.4 (SAS Institute, Cary, NC). Analysis of feasibility will be primarily descriptive. Numeric summaries including frequencies for categorical outcomes and means, medians, standard deviations and interquartile ranges for continuous outcomes will be presented. Graphical summaries will be used to describe distributions of outcomes and relations with baseline characteristics. 95% confidence intervals for means and proportions will be estimated to describe uncertainty from sampling variation for feasibility outcomes.

#2000031059

| 6.4.3.2 | Secondary | <b>Objectives</b> | Analyses |
|---------|-------------|-------------------|-----------|
| 0.4.3.2 | Secolidal v | ODIECTIVES | Allalvaca |

N/A

6.4.3.3 Safety

N/A

6.4.3.4 Analysis of Subject Characteristics

N/A

6.4.3.5 Interim Analysis (if applicable)

N/A

6.4.3.6 Health economic evaluation

N/A

6.4.3.7 Other

N/A

6.4.4 Subsets and Covariates

N/A

6.4.5 Handling of Missing Data

N/A

## 7 Trial Administration

#### 7.1 Ethical Considerations: Informed Consent/Assent and HIPAA Authorization

We pay special attention to the ethical issues and the unique challenges of EM research and to consenting and enrolling older adults in our study. We designed a detailed process on how to evaluate capacity, determine competence, and obtain informed consent from older adults. Evaluating the capacity of the participants to understand the purpose, risks, benefits, confidentiality, and privacy associated with the study is vital for valid informed consent. We will use standardized criteria to determine if the potential participant is capable of providing consent and by asking 2 questions: "What is the study about?" and "Can you stop the study at any time?".

Members of the study team who are responsible for participant recruitment and consent will be highly trained in obtaining informed consent. We will employ evidence-based practices from the geriatrics to correctly address these challenges. Evaluating the capacity of the participants to understand the purpose, risks, benefits, confidentiality, and privacy associated with study is vital for valid informed consent. Participants and/or LAR must be able to consent and communicate in English. The consent process will be done electronically, on the same tablet device as the VOICES tool. This electronic consent process was previously authorized for use with IRB #2000023799. Signed consent will be obtained and a print-out of the electronic text will be provided to the subject/LAR.

We are requesting a HIPPA waiver for recruitment purposes only. The RA will work with care team and will review the EPIC screen and will then check the demographic for patient 60 years or older. The YIMA staff will help the RA approach the patients to ask additional screening questions. We don't have resources and staffing to approach every **YIMA** patient and ascertain eligibility. Using Epic is more efficient for the RAs.

The RA will track and document each EHR that the RA accesses using the VOICES tool screening log.

1. What protected health information (medical information along with the HIPAA identifiers) about subjects will be collected and used for the research?

Medical records will be reviewed to collect the following variables: MRN, DOB, Able to communicate in English, Living in community dwelling, any severe hearing/vision impairment, and MoCA scores.

2. How will the research data be collected, recorded and stored?

We will have shadow files on each subject. Data of the study will be entered into a secure database. In this study, the following materials will be collected from human subjects: questionnaire, study subject's study ID, and signature. All paper documents will be maintained in a locked file, separate from other clinical records to assure confidentiality. All electronically stored data will be encrypted and password-protected. Only the primary investigator, co-investigators, study coordinator and programmers will have access to subjects' data. All datasets will be de-identified and only known to study investigators involved in consent and data acquisition. All information relating to participating subjects will be de-identified.

3. How will the digital data be stored?

On secure database server.

4. What methods and procedures will be used to safeguard the confidentiality and security of the identifiable study data and the storage media indicated above during and after the subject's participation in the study?

The VOICES system will be designed to ensure compliance with good research practice regarding the management of research data containing Protected Health Information (PHI). VOICES will adopt comprehensive security strategies that will assure the confidentiality and privacy of the patient and clinical information. Only authorized users will have access to patient PHI, which will help assuage concerns participants may have regarding the privacy and security of their data. The guidelines contained in the Common Framework give a detailed specification of technical architecture, privacy safeguards, and several approaches to health information exchange. We will utilize this framework to protect patient privacy and keep PHI under strict control. We will continuously evaluate our security practices in order to quickly identify any new vulnerabilities that could compromise VOICES integrity and privacy. We will utilize the Yale Information Technology Services (ITS) existing privacy and security practices and technology, and incorporate Yale ITS-consistent policies into VOICES development and implementation. In addition to tier separation and firewall protection, the system architecture maintains VOICES security, confidentiality, and privacy. VOICES will maintain data security with appropriate encryption, system controls and audit trails. Paper surveys will be stored in a locked area. All electronic data will be stored in secure database.

5. What will be done with the data when the research is completed? Are there plans to destroy the identifiable data? If yes, describe how, by whom and when identifiers will be destroyed. If no, describe how the data and/or identifiers will be secured.

Data will be stored in safe secure server.

6 If appropriate, has a Certificate of Confidentiality been obtained?

YES

### 7.2 Institutional Review Board (IRB) Review

The protocol will be submitted to the IRB for review and approval. Approval of the protocol must be obtained before initiating any research activity. Any change to the protocol or study team will require an approved IRB amendment before implementation.

A study closure report will be submitted to the IRB after all research activities have been completed.

Other study events (e.g. data breaches, protocol deviations) will be submitted per Yale IRB's policies.

#### 7.3 Subject Confidentiality

Subject confidentiality is held in strict trust by the research team. Subject medical record review will be limited to the just the elements needed to complete the study. Only authorized HIPAA and GCP trained study team members will be allowed to extract research data from medical records and enter it into VOICES database. No direct subject identifiers will be entered into VOICES data analysis database.

Each subject will be assigned a unique study number. A master list linking the unique study number to the human subject will be maintained in a secure database file.

#### 7.4 Deviations/Unanticipated Problems

If the study team becomes aware of an anticipated problem (e.g. data breach, protocol deviation), the event will be reported to the IRB by e-mail or via the IRES system as directed by the IRB.

#### 7.5 Data Collection

Data of the study will be entered into a secure database on a secure server. In this study, the following materials will be collected from human subjects: questionnaire, study subject's study ID, and signature. All paper documents will be maintained in a locked file, separate from other clinical records to assure confidentiality. All electronically stored data will be encrypted and password-protected. Only the primary investigator, co-investigators, study coordinator and programmers will have access to subjects' data. All datasets will be deidentified and only known to study investigators involved in consent and data acquisition. All information relating to participating subjects will be deidentified.

#### 7.6 Data Quality Assurance

The VOICES system will be designed to ensure compliance with good research practice regarding the management of research data containing Protected Health Information (PHI). VOICES will adopt comprehensive security strategies that will assure the confidentiality and privacy of the patient and clinical information. Only authorized users will have access to patient PHI, which will help assuage concerns participants may have regarding the privacy and security of their data. The guidelines contained in the Common Framework give a detailed specification of technical architecture, privacy safeguards, and several approaches to health information exchange. We will utilize this framework to protect patient privacy and keep PHI under strict local control. We will continuously evaluate our security practices in order to quickly identify any new vulnerabilities that could compromise VOICES integrity and privacy. We will utilize the Yale Information Technology Services (ITS) existing privacy and security practices and technology, and incorporate Yale ITS-consistent policies into VOICES development and implementation. In addition to tier separation and firewall protection, the three-tiered architecture maintains VOICES security, confidentiality, and privacy. VOICES will maintain data security with appropriate encryption, system controls and audit trails.

#### 7.7 Study Records

Documents that will be considered study records for this study are consent forms, demographics and post-use surveys.

#### 7.8 Access to Source

All documents will be collected electronically for the purpose of this study. All electronically stored data will be encrypted and password-protected. Only the primary investigator, co-investigators, study coordinator and programmers will have access to subjects' data. All datasets will be de-identified and only known to study investigators involved in consent and data acquisition.

#### 7.9 Data or Specimen Storage/Security

Data will be collected and stored digitally, and maintained on a securely encrypted database server with password protection.

#### 7.10 Retention of Records

Data will be retained based on Yale IRB policy.

#### 7.11 Study Monitoring

The Principal Investigator (PI) will be responsible for ensuring participants' safety on a daily basis.

#### 7.12 Data Safety Monitoring Plan

The DSMP will be monitored by the study team. The Principal Investigator (PI) will be responsible for ensuring participants' safety on a daily basis. To ensure that we are identifying both the adverse events that we might anticipate as well as those that we might not, the PI will review each case where either: (1) a report was made to PSE or (2) a patient was admitted to the hospital for safety to assess for any potential adverse events. The Data and Safety Monitoring Team (DSMT) will consist of Drs. Abujarad, Hwang, and Marottoli; this team will monitor participant safety, evaluate the progress of the study, and review procedures for maintaining the confidentiality of data, the quality of data collection, management, and analyses. They will monitor the study for reports of any adverse or unexpected events. Study participants will be advised to contact the study team to report any adverse events or concerns. VOICES will only be administrated for the intervention group, and there will be no control groups. The PI and the investigative team will monitor data and safety at the monthly study team meetings.

The following will be reviewed:

- Cumulative accrual
- Enrollment of subjects who meet the study eligibility criteria only
- Recruitment is proceeding as planned
- The informed consent process is conducted appropriately; informed consent is obtained
- Evaluate the progress of the trial, including periodic assessments of data quality and timeliness, recruitment, accrual and retention, participant risk versus benefit, and other factors that can affect study outcome
- Consider factors external to the study when relevant information becomes available, such as scientific or therapeutic developments that may have an impact on the safety of the participants or the ethics of the trial
- Review study performance, make recommendations, and assist in the resolution of problems reported by the PI
- Evaluate data completeness and quality and as specified in the protocol

Prior to proceeding with any study procedures:

- Review the research protocol, informed consent documents and plans for data safety and monitoring
- Protect the safety of the study participants
- Ensure the confidentiality of the study data and the results of monitoring
- Review procedures for the privacy and confidentiality of subjects
- Review cumulative attrition and attrition by gender and race/ethnicity
- Review dropouts and ensure reason for withdrawal from the study are documented

The principal investigator will be responsible for monitoring the data, assuring protocol compliance, and conducting the safety reviews. During the review process the principal investigator will evaluate whether the study should continue unchanged, require modification/amendment, or close enrollment. The principal investigator and the

Institutional Review Board (IRB) and the NIA have the authority to stop or suspend the study or require modifications.

## 7.13 Study Modification

For any study modifications, we will update this study protocol. Then we will submit the updated protocol to Yale IRB for approval. Once approved the changes can be implemented in the study.

#### 7.14 Study Discontinuation

N/A

#### 7.15 Study Completion

The study will be completed by December 31<sup>th</sup> 2022. The PI will notify Yale IRB of the study completion.

## 7.16 Conflict of Interest Policy

The independence of this study from any actual or perceived influence, such as by the pharmaceutical industry, is critical. Therefore, any actual conflict of interest of persons who have a role in the design, conduct, analysis, publication, or any aspect of this trial will be disclosed and managed. Furthermore, persons who have a perceived conflict of interest will be required to have such conflicts managed in a way that is appropriate to their participation in the trial. The study leadership in conjunction with the appropriate conflict of interest review committee has established policies and procedures for all study group members to disclose all conflicts of interest and will establish a mechanism for the management of all reported dualities of interest.

All investigators will follow the applicable conflict of interest policies.

## 7.17 Funding Source

The study is funded by the Yale Claude D. Pepper Older Americans Independence Center OAIC Sponsor Award (IRES #: 18-001844-011).

#### 7.18 Publication Plan

At the completion of this study and the feasibility study for older adults with cognitive impairment, we expect to enhance the VOICES tool and create all related and necessary user guides. We anticipate that if feasible, VOICES will inform development of national Elder Mistreatment (EM) intervention and screening guidelines on a generalizable scale that will broaden the base for EM identification and intervention while closing health disparity gaps and respecting the autonomy of older adults. Yale University is committed to open and timely dissemination of research outcomes and is aware of and agrees to abide by the principles for sharing research resources.

#2000031059

# 8 Appendices

| Appendix # Title | Section | Topic |
|------------------|---------|-------|
|------------------|---------|-------|

#2000031059

01/20/22 Version #1.01

# 9 List of Tables